CLINICAL TRIAL: NCT01384357
Title: Real-time Ultrasound-Guided Needle Biopsy in the Diagnosis of Malignant Cervical Lymphadenopathies
Brief Title: Ultrasound-Guided Needle Biopsy in the Diagnosis of Malignant Cervical Lymphadenopathies
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Liao Li-Jen, Department of Otolaryngology, Far Eastern Memorial Hospital
Other Study IDs: 100026-E
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-05

CONDITIONS: Lymphadenopathy; Malignancy
Keywords: lymphadenopathy; needle biopsy; sonography
MeSH Terms: conditions — Lymphadenopathy; Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ultrasound,lymphadenopathy

SUMMARY:
The objective of the present study was to compare ultrasound (US) characteristics and ultrasound-guided core-needle biopsy (US-CNB) with US-guided fine-needle aspiration (US-FNA) in the assessment of different malignant cervical lymphadenopathies. Patients with malignant cervical lymphadenopathie with either US-FNA or US-CNB over a 3-year period from 2007 July to 2010 Dec were retrospectively reviewed. There are two major study groups according to the treatment status of the patient's population, including patients who had pathology proofed previous cancer and with clinically cervical lymphadenopathies after treatment. The second group included patients with cervical lymphaenopathies but without previous diagnosis of malignancy and treatment. The results of cytology, or pathology and time of needle biopsy to final diagnosis were traced and recorded. Morphologic US parameters and vascular features were thoroughly evaluated and compared in different disease.

DETAILED DESCRIPTION:
Introduction

In the absence of infection signs, lateral neck lymphadenopathies should be suspected as metastatic carcinoma or lymphoma until proved otherwise. Previously, the most commonly used sampling techniques in the head and neck are the open excisional biopsy and fine-needle aspiration (FNA) cytology. Open biopsy and lymph node excision provides material suitable for histological analysis but is invasive and may entail general anesthesia and hospital admission. Besides, excisional and incisional biopsy of cervical metastases results in a 2-3 times increased incidence of local treatment failure when compared with FNA cytology.

High-resolution ultrasound is widely used imaging modality to evaluate the morphology, internal architecture, size and shape of cervical lymph nodes. In the head and neck, the image guidance technique most commonly used has been ultrasound. The real-time capability and ease of use makes ultrasound the procedure of choice. The evidence of improved efficacy of ultrasound-guided FNA over palpation-guided FNA in the head and neck also has been well documented, leading to its acceptance as the standard procedure.

Disadvantages of FNA include a high rate of nondiagnostic samples and incomplete classification of lymphoma with delayed diagnosis. The core-needle biopsy (CNB) is an alternative to the established ways of tissue sampling and used very successfully for many years. As the histologic architecture of the lesion is preserved, it provides a sample that is adequate for histopathologic and immunohistochemical examination.

To our knowledge, there was only one prospective investigation comparing ultrasound guided CNB with FNA in the head and neck region. However, the studied population was heterogeneous and case numbers were limited. The result revealed no significant difference between both methods. The objective of the present study was to compare ultrasound-guided CNB with FNA in the assessment of different malignant cervical lymphadenopathies.

Patients and methods

A retrospective study will be performed including consecutive patients over a 3-year period from 2007 July to 2010 Dec. All patients were seen at our institution with malignant cervical lymphadenopathies. The biopsies were performed on an outpatient basis, unless the patient was hospitalized for alternative reasons. Equipment for sonographic studies consisted of a color Doppler US unit (Philips HDI 5000, Bothell, WA, US) and a 5-12 MHz broadband linear array transducer.

Morphologic US parameters and vascular features were thoroughly evaluated and recorded on the PACS system (Marotech Inc, Seoul, South Korea) for the largest nodal lesion in each patient. Every lymph node was assessed first with gray-scale sonography for morphologic parameters in horizontal and then longitudinal sections. The short-axis diameter, long-axis diameter and diameter ratio of short to long axis (S/L ratio) were measured. Echogenicity with respect to the surrounding soft tissue was assessed and classified as hypoechoic, isoechoic, or hyperechoic. Lymph node margin was defined as regular or irregular. Echogenic hilus was distinguished between its presence or absence. Internal echo pattern was divided into heterogeneity or homogeneity. Vascular patterns were then surveyed by power Doppler sonography and categorized as the group of avascular or hilar type versus that of mixed, spotted, or peripheral type.

With the data on history, physical examination, and ultrasound result, we decided that ultrasound guided needle biopsies would be the first line of investigation for these lesions. Informed consent for the procedure was obtained from all the patients before biopsy. In general, FNA was carried out with the array probe guiding the placement of a 22-gauge fine needle within the largest node after sterilization without anesthesia. For CNB, the skin was sterilized and locally anaesthetized with 2% lidocaine. A modified non-advancing, disposable, spring-loaded cutting biopsy needle (Temno biopsy system, Allegiance Healthcare Corporation, McGaw Park, IL, USA) with 15-mm side-notch of 9 cm length and 18-gauge were used. All biopsies were done by the same experienced otolaryngologist (Li-Jen Liao) under real-time ultrasound guidance with freehand technique. Three times of tissue core biopsies were done for each patient. After the biopsy, all patients were asked to compress the puncture site and were evaluated for possible complications such as bleeding or bruising for half an hour before leaving the examination room.

The specimens were put in 10% formalin solution for pathologic studies. In the Department of Pathology, formalin-fixed, paraffin-embeddedm sections from the biopsies were stained with hematoxylin and eosin for morphologic examination. Further immunohistochemical studies were performed as necessary.

There are two major study groups according to the treatment status of the patient's population. The first group included patients who had pathology proofed previous cancer and with clinically cervical lymphadenopathies after treatment. The second group included patients with cervical lymphaenopathies but without previous diagnosis of malignancy and treatment. The disease groups were further classified as metastatic nodes from nonthyroid primary (META), lymphoma (LYM) and metastatic nodes from papillary carcinoma of the thyroid (PAP).

The results of cytology and pathology were graded as false negative, suspicious and positive for malignancy. The final diagnoses of patients were established by the histopathology. The time of needle biopsy and final diagnosis were traced and recorded.

Statistically, continuous variables were compared by performing the Kruskal-Wallis test. Category data were compared by using the Chi-square test or Fisher's exact test. The time from procedure to final diagnosis were expressed in K-M plot and tested with Log-rank test. All statistical analyses were accomplished using SAS software, version 9.1 (SAS Institute, Inc, Cary, North Carolina).

Expected Results:

We will know the differential US characteristics in different malignant cervical lymphadenopathies. Besides, we will know US-FNA or US-CNB is preferred in which situation.

ELIGIBILITY:
Inclusion Criteria:

Patients with malignant cervical lymphadenopathie With US-FNA or US-CNB evaluation before

Exclusion Criteria:

No ultrasound exam

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant cervical lymphadenopathie with either US-FNA or US-CNB over a 3-year period from 2007 July to 2010 Dec were retrospectively reviewed. There are two major study groups according to the treatment status of the patient's population, including patients who had pathology proofed previous cancer and with clinically cervical lymphadenopathies after treatment. The second group included patients with cervical lymphaenopathies but without previous diagnosis of malignancy and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2007-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
time of needle biopsy to final diagnosis | days from needle biopsy to final diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jen Liao, M.D., Principal Investigator — Department of Otolaryngology, Far Eastern Memorial Hospital, New Taipei City, Taiwan
Locations (1):
- Department of Otolaryngology, Far Eastern Memorial Hospital, Taipei, Taiwan